CLINICAL TRIAL: NCT01469793
Title: A Phase I, Open Label Study of the Safety and Pharmacokinetics of Escalating Doses of DMOT4039A in Patients With Unresectable Pancreatic or Platinum-Resistant Ovarian Cancer
Brief Title: A Study of DMOT4039A in Participants With Unresectable Pancreatic or Platinum-Resistant Ovarian Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DMO4993g; GP27896 (Other: Hoffmann-La Roche); 2011-002713-10 (EudraCT Number)
Record Dates: First submitted 2011-11-07; First posted 2011-11-10 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2016-11

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

ARMS (4):
- DMOT4039A Q3W: Dose Escalation (Experimental): Participants in different cohorts will receive DMOT4039A at various escalating dose levels, starting with 0.2 milligrams per kilogram (mg/kg), as intravenous infusion every 3 weeks (Q3W) to determine the maximum tolerated dose (MTD) of DMOT4039A for until disease progression, loss of clinical benefit or unacceptable toxicity, whichever occurred first (up to approximately 2.5 years).
  Interventions: Drug: DMOT4039A
- DMOT4039A Q3W: Dose Expansion (Experimental): Participants will receive DMOT4039A at recommended phase 2 dose (RP2D) for Q3W dosing schedule as intravenous infusion Q3W until disease progression, loss of clinical benefit or unacceptable toxicity, whichever occurred first (up to approximately 2.5 years).
  Interventions: Drug: DMOT4039A
- DMOT4039A Q1W: Dose Escalation (Experimental): Participants in different cohorts will receive DMOT4039A at various escalating dose levels, starting with a dose 33% of MTD for Q3W dosing schedule, as intravenous infusion every week (Q1W) to determine the MTD of DMOT4039A for until disease progression, loss of clinical benefit or unacceptable toxicity, whichever occurred first (up to approximately 2.5 years).
  Interventions: Drug: DMOT4039A
- DMOT4039A Q1W: Dose Expansion (Experimental): Participants will receive DMOT4039A at RP2D for Q1W dosing schedule as intravenous infusion Q1W until disease progression, loss of clinical benefit or unacceptable toxicity, whichever occurred first (up to approximately 2.5 years).
  Interventions: Drug: DMOT4039A

INTERVENTIONS:
Drug: DMOT4039A — DMOT4093A will be administered by intravenous infusion on either a Q3W or a Q1W dosing schedule, in 21-day cycles.

SUMMARY:
This multicenter, open-label, dose-escalating study will assess the safety, tolerability, and pharmacokinetics of DMOT4039A in participants with unresectable pancreatic or platinum-resistant ovarian cancer. Cohorts of participants will receive multiple ascending intravenous doses of DMOT4039A.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Histologically documented, incurable, locally advanced or metastatic disease for which no standard therapy exists, consisting of one of the following: Unresectable pancreatic ductal adenocarcinoma or platinum-resistant ovarian cancer
* Measureable disease, defined as at least one bi-dimensionally measurable non-lymph node lesion greater than or equal to (>/=) 1 centimeter (cm) in long-axis diameter on spiral computed tomography (CT) scan or at least one bi-dimensionally measurable lymph node measuring >/= 1.5 cm in short-axis diameter on spiral CT scan
* Adequate hematological, renal and liver function

Exclusion Criteria:

* Treatment with anti-tumor therapy, including chemotherapy, biologic, experimental or hormonal therapy, within 4 weeks prior to Day 1
* Known active infection
* Current Grade >/= 2 toxicity (except for alopecia, anorexia and fatigue) from prior therapy or Grade >/= 2 neuropathy
* Untreated or active cerebral nervous system metastases
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2011-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of DMOT4039A | Days 1 to 21 of Cycle 1 (1 cycle=21 days)
Number of Participants With Dose-Limiting Toxicities (DLTs) | Days 1 to 21 of Cycle 1 (1 cycle=21 days)
Recommended Phase 2 Dose (RP2D) of DMOT4039A | Days 1 to 21 of Cycle 1 (1 cycle=21 days)

SECONDARY OUTCOMES:
Area Under the Concentration-Time Curve From Time Zero to Extrapolated Infinite Time (AUC [0-inf]) of DMOT4039A Total Antibody | Q3W: Pre-infusion (0 hours [hrs]), 0.5, 4, 24, 48 hrs, and 7, 9/10, 14, 16/17 days post-infusion in Cycle 1; Q1W: Pre-infusion, 0.5, 48 hrs post Day 1, 8, 15 infusions, 4, 24 hrs post Day 1 infusion in Cycle 1 (Infusion length=1.5 hrs) (1 cycle=21 days)
AUC (0-inf) of Antibody-Conjugated Monomethyl Auristatin E (acMMAE) | Q3W: Pre-infusion (0 hrs), 0.5, 4, 24, 48 hrs, and 7, 9/10, 14, 16/17 days post-infusion in Cycle 1; Q1W: Pre-infusion (0 hrs), 0.5, 48 hrs post Day 1, 8, 15 infusions, 4, 24 hrs post Day 1 infusion in Cycle 1 (Infusion length=1.5 hrs) (1 cycle=21 days)
AUC (0-inf) of Unconjugated MMAE | Q3W: Pre-infusion (0 hrs), 0.5, 4, 24, 48 hrs, and 7, 9/10, 14, 16/17 days post-infusion in Cycle 1; Q1W: Pre-infusion (0 hrs), 0.5, 48 hrs post Day 1, 8, 15 infusions, 4, 24 hrs post Day 1 infusion in Cycle 1 (Infusion length=1.5 hrs) (1 cycle=21 days)
Maximum Observed Concentration (Cmax) of DMOT4039A Total Antibody | Q3W: Pre-infusion (0 hrs), 0.5, 4, 24, 48 hrs, and 7, 9/10, 14, 16/17 days post-infusion in Cycle 1; Q1W: Pre-infusion (0 hrs), 0.5, 48 hrs post Day 1, 8, 15 infusions, 4, 24 hrs post Day 1 infusion in Cycle 1 (Infusion length=1.5 hrs) (1 cycle=21 days)
Cmax of acMMAE | Q3W: Pre-infusion (0 hrs), 0.5, 4, 24, 48 hrs, and 7, 9/10, 14, 16/17 days post-infusion in Cycle 1; Q1W: Pre-infusion (0 hrs), 0.5, 48 hrs post Day 1, 8, 15 infusions, 4, 24 hrs post Day 1 infusion in Cycle 1 (Infusion length=1.5 hrs) (1 cycle=21 days)
Cmax of Unconjugated MMAE | Q3W: Pre-infusion (0 hrs), 0.5, 4, 24, 48 hrs, and 7, 9/10, 14, 16/17 days post-infusion in Cycle 1; Q1W: Pre-infusion (0 hrs), 0.5, 48 hrs post Day 1, 8, 15 infusions, 4, 24 hrs post Day 1 infusion in Cycle 1 (Infusion length=1.5 hrs) (1 cycle=21 days)
Total Clearance (CL) of DMOT4039A Total Antibody | Q3W: Pre-infusion (0 hrs), 0.5, 4, 24, 48 hrs, and 7, 9/10, 14, 16/17 days post-infusion in Cycle 1; Q1W: Pre-infusion (0 hrs), 0.5, 48 hrs post Day 1, 8, 15 infusions, 4, 24 hrs post Day 1 infusion in Cycle 1 (Infusion length=1.5 hrs) (1 cycle=21 days)
CL of acMMAE | Q3W: Pre-infusion (0 hrs), 0.5, 4, 24, 48 hrs, and 7, 9/10, 14, 16/17 days post-infusion in Cycle 1; Q1W: Pre-infusion (0 hrs), 0.5, 48 hrs post Day 1, 8, 15 infusions, 4, 24 hrs post Day 1 infusion in Cycle 1 (Infusion length=1.5 hrs) (1 cycle=21 days)
Half-life (t1/2) of DMOT4039A Total Antibody | Q3W: Pre-infusion (0 hrs), 0.5, 4, 24, 48 hrs, and 7, 9/10, 14, 16/17 days post-infusion in Cycle 1; Q1W: Pre-infusion (0 hrs), 0.5, 48 hrs post Day 1, 8, 15 infusions, 4, 24 hrs post Day 1 infusion in Cycle 1 (Infusion length=1.5 hrs) (1 cycle=21 days)
t1/2 of acMMAE | Q3W: Pre-infusion (0 hrs), 0.5, 4, 24, 48 hrs, and 7, 9/10, 14, 16/17 days post-infusion in Cycle 1; Q1W: Pre-infusion (0 hrs), 0.5, 48 hrs post Day 1, 8, 15 infusions, 4, 24 hrs post Day 1 infusion in Cycle 1 (Infusion length=1.5 hrs) (1 cycle=21 days)
t1/2 of Unconjugated MMAE | Q3W: Pre-infusion (0 hrs), 0.5, 4, 24, 48 hrs, and 7, 9/10, 14, 16/17 days post-infusion in Cycle 1; Q1W: Pre-infusion (0 hrs), 0.5, 48 hrs post Day 1, 8, 15 infusions, 4, 24 hrs post Day 1 infusion in Cycle 1 (Infusion length=1.5 hrs) (1 cycle=21 days)
Volume of Distribution at Steady State (Vss) of DMOT4039A Total Antibody | Q3W: Pre-infusion (0 hrs), 0.5, 4, 24, 48 hrs, and 7, 9/10, 14, 16/17 days post-infusion in Cycle 1; Q1W: Pre-infusion (0 hrs), 0.5, 48 hrs post Day 1, 8, 15 infusions, 4, 24 hrs post Day 1 infusion in Cycle 1 (Infusion length=1.5 hrs) (1 cycle=21 days)
Vss of acMMAE | Q3W: Pre-infusion (0 hrs), 0.5, 4, 24, 48 hrs, and 7, 9/10, 14, 16/17 days post-infusion in Cycle 1; Q1W: Pre-infusion (0 hrs), 0.5, 48 hrs post Day 1, 8, 15 infusions, 4, 24 hrs post Day 1 infusion in Cycle 1 (Infusion length=1.5 hrs) (1 cycle=21 days)
Percentage of Participants With Anti-Therapeutic Antibodies (ATAs) | Baseline (pre-infusion [0 hrs] on Day 1 Cycle 1); Post-Baseline (assessed at pre-infusion [0 hrs] on Day 1 of Cycles 2-4 and at study completion/early termination [up to 30 days after Cycle 32]) (1 cycle=21 days)
Percentage of Participants With Objective Response According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) | Baseline up to PD or death, whichever occurred first (assessed at Day 1, every 2 cycles thereafter [Cycles 2, 4, 6, 8, 10, 12, 14, and 16]; at study completion/early withdrawal [up to 30 days after Cycle 32]) (1 cycle=21 days)
Duration of Objective Response (DOR) According to RECIST v1.1 | From the date of initial PR or CR up to PD or death, whichever occurred first (assessed at Day 1, every 2 cycles thereafter [Cycles 2, 4, 6, 8, 10, 12, 14, and 16]; at study completion/early withdrawal [up to 30 days after Cycle 32]) (1 cycle=21 days)
Progression-free Survival (PFS) According to RECIST v1.1 | Day 1 up to PD or death, whichever occurred first (assessed at Day 1, every 2 cycles thereafter [Cycles 2, 4, 6, 8, 10, 12, 14, and 16]; at study completion/early withdrawal [up 30 days after Cycle 32]) (1 cycle=21 days)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (6):
- United States (4):
  - Phoenix, Arizona
  - Aurora, Colorado
  - Jacksonville, Florida
  - Rochester, Minnesota
- Netherlands (2):
  - Amsterdam
  - Groningen